CLINICAL TRIAL: NCT03069222
Title: Longitudinal Assessment of Spinal Cord Structural Plasticity Using DTI in SCI Patients
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Bing Yao, PhD, Senior Physicist and Manager, Kessler Foundation
Other Study IDs: Kessler
Record Dates: First submitted 2017-02-14; First posted 2017-03-03 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injuries
Keywords: diffusion tensor imaging
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: SCI patients enrolled at Kessler Institute Rehabiliation
  Interventions: Other: Standard Rehabilitative Treatment
- Control: age and gender matched with patient enrolled

INTERVENTIONS:
Other: Standard Rehabilitative Treatment — The patients will participate in standard but comprehensive SCI specific rehabilitation therapy provided by the SCI program at KIR. The therapy consists of 3 hours per day, 5 days a week. Motor function therapy includes standardized procedures for range of motion, passive and active muscle activities, and therapies to improve mobility. The treatment program for the enrolled patients will be standardized by Dr. Kirshblum, Director of the SCI program at KIR and a Co-Investigator of the study. Patients usually receive 4 weeks of rehabilitation treatment; however, if any of them are discharged earlier from KIR, their out-patient treatment activities will be monitored and the patients will be tested based on the planned schedule.
  Groups: Patient

SUMMARY:
This study will apply novel magnetic resonance imaging (MRI) techniques to investigation of spinal cord injury (SCI) to learn how nerve fibers repair and neural cells regain ability to control muscle during the rehabilitation. The information gained will be helpful for physicians to make more accurate diagnosis of SCI, predict injury recovery and movement restoration, and develop more effective treatment plans.

DETAILED DESCRIPTION:
Today, the International Standards for the Neurological Classification of Spinal Cord Injury (ISNSCI) , which includes tests of motor and cutaneous sensory function, and Spinal Cord Independence Measure (SCIM) are the gold standards for neurological classification of spinal cord injury (SCI). These standard measures have very important applications in the rehabilitation of SCI as primary clinical and outcome measures. Despite the importance and usefulness of their applications, these standard measures have their limitations. For example, ISNSCI, intended to be a clinical classification system, is subjective and relatively insensitive to incremental neurophysiological and functional changes during both acute and chronic stages of recovery. Moreover, the ISNSCI cannot evaluate the spinal cord (SC) function bellow the neurological level. For some patients such as children and patients with concomitant brain injuries, reliable evaluation cannot be completed due to their limited cognitive engagement in the evaluation process. Magnetic resonance imaging (MRI) has been proposed as a more objective tool to help clinicians make prognosis. However, recent study showed that conventional clinical MRI does not correlate well with scores measured with ISNSCI.

Diffusion Tensor Imaging (DTI) is an advanced MRI tool capable of probing white matter integrity information through measuring directional diffusion of water molecules, thus providing more microscopic details than conventional MRI. Recent findings suggest that DTI is a promising, non-invasive and objective tool for evaluating and monitoring structural changes within white matter axon pathways after SCI. Our preliminary data showed significant deviation of DTI indices from normative values of healthy subjects in a SCI patient whose conventional T2 scans appeared to be normal (see preliminary data section). A likely explanation for this observed alteration of DTI indices is degeneration and demyelization in descending axonal pathways. Although DTI has been used in animal models to measure the evolution of the injury in the SC and showed great promise in detection of pathological changes in SC, no longitudinal DTI data obtained from human SC are available to indicate sensitivity of DTI technique in detecting SCI progression or recovery. Is DTI capable of detecting structural changes taking place in the SC over the course of rehabilitation in individuals with SCI? Will these measured DTI parameters correlate with ISNSCI-based scores? The fundamental hypothesis of the current study is that rehabilitation can facilitate SC fiber tract repair along with spontaneous adaptations following the injury to help reconnect some of the injured nerve fibers with motoneurons controlling muscles and this will in turn improve the motoneuron activity to promote muscular function, and all these changes can be detected by the proposed longitudinal DTI protocols and standard clinical tools for motor function evaluation. The expected results gained by this longitudinal study would support the application of DTI in monitoring plastic changes in the injured SC and the DTI-derived measures could potentially aid clinicians make more objective diagnosis of the injury and estimate its progression, which are critical in planning targeted therapies. However, it is out of the scope of this proposal to distinguish contributions to structural changes occurring in the SC between spontaneous and treatment factors. Because it is unethical to not treat patients, this limitation cannot be overcome in the current human study. Given the primary focus of the study being longitudinal tracking of SC structural changes using neuroimaging rather than determining relative contributions to these changes by spontaneous recovery and treatment, the limitation should not significantly influence the quality of our study. To test the hypothesis, the investigators propose the following Specific Aims.

Aim 1: Track SC structural changes in patients with incomplete SCI (iSCI) using DTI. Each patient in the proposed study will be scanned covering entire cervical region of the SC using a DTI sequence at baseline, 2 weeks, 1 month, 3 month and 6 month after start of standard rehabilitation intervention. DTI indices (see methods for details) will be quantified and compared across all time points. Previous longitudinal brain DTI human and animal studies suggest that DTI is sensitive to detect brain whiter matter structural changes 24 hours (animal study) and 3 months (unpublished human DTI results by PI's group) after brain injury, and 6 month after initial scan in patients with Amyotrophic lateral sclerosis(ALS) (DTI data were only available 6 months after initial scan in this study). The investigators hypothesize that the proposed DTI protocol will be able to capture structural changes in SCI during its recovery course.

Aim 2: Correlate the SC plasticity manifested by changes in DTI indices with clinical assessments of injury and sensorimotor function. Quantitative DTI indices will be correlated to clinical diagnoses of SCI and clinical evaluations of upper and lower limb sensorimotor function of the patients. It is hypothesized that the DTI index of SCI will significantly be correlated with clinical diagnosis and scores of upper and lower sensorimotor function. The DTI parameter holds great promise to be a biomarker of SCI and is expected to have prognostic value in predicting functional outcome of a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* SCI due to single event traumatic injury; C4-T12 neurological level of injury, AIS grade B,C or D;
* currently medically stable;
* no history of seizure;
* spasticity at a score of 2 or lower assessed using Modified Ashworth Assessment of the upper and lower extremities;
* able to give informed consent;
* to stay still in the MR scanner for ~30 min.

Exclusion Criteria:

* MRI contraindications;
* younger than 18 and older than 75 years (this age range will limit contributions from nervous system development and aging to results of the study);
* history of epilepsy and other neurological diseases and trauma;
* drug and alcohol abuse;
* multi injury levels;
* severe craniocerebral injury and
* presence of non-MRI-safe post-operative hardware in the spine or brain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twelve (12) individuals with iSCI (within 3 weeks post injury) will be recruited from Kessler Institute for Rehabilitation (KIR). In addition, we will recruit twelve healthy age- and gender-matched controls. All participants will give informed consent. For the SCI group the following clinical evaluations will occur at baseline, 2 weeks, 1 month, 3 months and 6 months by the study physician or clinician.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | changes within 6 months after participant enrolls.
  Neurological examination will be performed using the ISNCSCI. Sensory scores and lower and upper extremity motor scores (LEMS and UEMS) are derived at the time of this exam. The ISNCSCI and all examinations described below will be performed following the same schedule as the imaging (DTI, T2, T2*) evaluation (baseline, 2 weeks, 1 month, 3 months, and 6 months after commencement of rehabilitation therapy). The LEMS measures strength in five muscle groups bilaterally (hip flexors, knee flexors, extensors, and ankle dorsiflexors) and the UEMS also assess strength bilaterally in 5 muscle groups (elbow flexors, elbow extensors, wrist extensors, finger flexors, finger abductors) with the modified British Medical Research Council scale and is performed during the ISNCSCI examination.
Modified Ashworth Scale (MAS) | changes within 6 months after participant enrolls.
  Spasticity assessments will be performed at each visit using the MAS. It tests the resistance to passive movement about a joint with vary degrees of velocity. The scores range from 0 to 4, with 6 choices (0, 1, 1+, 2, 3, and 4). A score of 0 indicates no resistance, and 4 indicates rigidity. The MAS scores will be averaged across 5 muscle groups bilaterally for lower extremities and 5 muscle groups for upper extremities. An experienced therapist will perform all the evaluations for all the visits and all subjects.
Spinal Cord Independence measure III (SCIM III) | changes within 6 months after participant enrolls.
  The SCIM is a measure of functional ability developed specifically for individuals with SCI to evaluate their performance of activities of daily living and to make functional assessments of this population sensitive to change. SCIM scores a task higher in patients who accomplish it with less assistannce, aids, or medical compromise than other patients. The SCIM III to be adopted by the current study is composed of 19 items in 3 subscales: (a) self-care; (b) respiration and sphincter management; and (c) mobility. The total score ranges from 0 to 100. Mobility is subdivided into "room and toilet" and "indoors and outdoors". The items are weighted in terms of their assumed clinical relevance. The SCIM III is a valid and reliable measure and is recommended as a primary outcome measure to assess functional recovery in individuals with SCI.

SECONDARY OUTCOMES:
Diffusion Tensor Image | before [baseline] and 2 weeks, 1 month, 3 months and 6 months after commencement of rehabilitative treatment)
  Being an advanced MRI tool, DTI provides excellent structural information on microscopic level such as remyelination which plays an important role in rehabilitation of SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Yao, Ph.D., Principal Investigator — Kessler Fondation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirshblum SC, Waring W, Biering-Sorensen F, Burns SP, Johansen M, Schmidt-Read M, Donovan W, Graves D, Jha A, Jones L, Mulcahey MJ, Krassioukov A. Reference for the 2011 revision of the International Standards for Neurological Classification of Spinal Cord Injury. J Spinal Cord Med. 2011 Nov;34(6):547-54. doi: 10.1179/107902611X13186000420242. PMID 22330109
- [Background] Marino RJ, Graves DE. Metric properties of the ASIA motor score: subscales improve correlation with functional activities. Arch Phys Med Rehabil. 2004 Nov;85(11):1804-10. doi: 10.1016/j.apmr.2004.04.026. PMID 15520975
- [Background] Mulcahey MJ, Samdani AF, Gaughan JP, Barakat N, Faro S, Shah P, Betz RR, Mohamed FB. Diagnostic accuracy of diffusion tensor imaging for pediatric cervical spinal cord injury. Spinal Cord. 2013 Jul;51(7):532-7. doi: 10.1038/sc.2013.36. Epub 2013 Apr 23. PMID 23608812
- [Background] Chang Y, Jung TD, Yoo DS, Hyun JK. Diffusion tensor imaging and fiber tractography of patients with cervical spinal cord injury. J Neurotrauma. 2010 Nov;27(11):2033-40. doi: 10.1089/neu.2009.1265. PMID 20822462
- [Background] Cheran S, Shanmuganathan K, Zhuo J, Mirvis SE, Aarabi B, Alexander MT, Gullapalli RP. Correlation of MR diffusion tensor imaging parameters with ASIA motor scores in hemorrhagic and nonhemorrhagic acute spinal cord injury. J Neurotrauma. 2011 Sep;28(9):1881-92. doi: 10.1089/neu.2010.1741. Epub 2011 Aug 29. PMID 21875333
- [Background] Toma K, Matsuoka T, Immisch I, Mima T, Waldvogel D, Koshy B, Hanakawa T, Shill H, Hallett M. Generators of movement-related cortical potentials: fMRI-constrained EEG dipole source analysis. Neuroimage. 2002 Sep;17(1):161-73. doi: 10.1006/nimg.2002.1165. PMID 12482074
- [Background] Freund P, Curt A, Friston K, Thompson A. Tracking changes following spinal cord injury: insights from neuroimaging. Neuroscientist. 2013 Apr;19(2):116-28. doi: 10.1177/1073858412449192. Epub 2012 Jun 22. PMID 22730072
- [Background] Brennan FH, Cowin GJ, Kurniawan ND, Ruitenberg MJ. Longitudinal assessment of white matter pathology in the injured mouse spinal cord through ultra-high field (16.4 T) in vivo diffusion tensor imaging. Neuroimage. 2013 Nov 15;82:574-85. doi: 10.1016/j.neuroimage.2013.06.019. Epub 2013 Jun 14. PMID 23770410
- [Background] Keil C, Prell T, Peschel T, Hartung V, Dengler R, Grosskreutz J. Longitudinal diffusion tensor imaging in amyotrophic lateral sclerosis. BMC Neurosci. 2012 Nov 8;13:141. doi: 10.1186/1471-2202-13-141. PMID 23134591
- [Background] Mac Donald CL, Dikranian K, Song SK, Bayly PV, Holtzman DM, Brody DL. Detection of traumatic axonal injury with diffusion tensor imaging in a mouse model of traumatic brain injury. Exp Neurol. 2007 May;205(1):116-31. doi: 10.1016/j.expneurol.2007.01.035. Epub 2007 Feb 12. PMID 17368446
- [Background] Koskinen E, Brander A, Hakulinen U, Luoto T, Helminen M, Ylinen A, Ohman J. Assessing the state of chronic spinal cord injury using diffusion tensor imaging. J Neurotrauma. 2013 Sep 15;30(18):1587-95. doi: 10.1089/neu.2013.2943. Epub 2013 Aug 9. PMID 23758292
- [Background] ASHWORTH B. PRELIMINARY TRIAL OF CARISOPRODOL IN MULTIPLE SCLEROSIS. Practitioner. 1964 Apr;192:540-2. No abstract available. PMID 14143329
- [Background] Kirshblum S, Millis S, McKinley W, Tulsky D. Late neurologic recovery after traumatic spinal cord injury. Arch Phys Med Rehabil. 2004 Nov;85(11):1811-7. doi: 10.1016/j.apmr.2004.03.015. PMID 15520976
- [Background] Anderson K, Aito S, Atkins M, Biering-Sorensen F, Charlifue S, Curt A, Ditunno J, Glass C, Marino R, Marshall R, Mulcahey MJ, Post M, Savic G, Scivoletto G, Catz A; Functional Recovery Outcome Measures Work Group. Functional recovery measures for spinal cord injury: an evidence-based review for clinical practice and research. J Spinal Cord Med. 2008;31(2):133-44. doi: 10.1080/10790268.2008.11760704. PMID 18581660
- [Background] Catz A, Itzkovich M, Tesio L, Biering-Sorensen F, Weeks C, Laramee MT, Craven BC, Tonack M, Hitzig SL, Glaser E, Zeilig G, Aito S, Scivoletto G, Mecci M, Chadwick RJ, El Masry WS, Osman A, Glass CA, Silva P, Soni BM, Gardner BP, Savic G, Bergstrom EM, Bluvshtein V, Ronen J. A multicenter international study on the Spinal Cord Independence Measure, version III: Rasch psychometric validation. Spinal Cord. 2007 Apr;45(4):275-91. doi: 10.1038/sj.sc.3101960. Epub 2006 Aug 15. PMID 16909143
- [Background] Anderson KD, Acuff ME, Arp BG, Backus D, Chun S, Fisher K, Fjerstad JE, Graves DE, Greenwald K, Groah SL, Harkema SJ, Horton JA 3rd, Huang MN, Jennings M, Kelley KS, Kessler SM, Kirshblum S, Koltenuk S, Linke M, Ljungberg I, Nagy J, Nicolini L, Roach MJ, Salles S, Scelza WM, Read MS, Reeves RK, Scott MD, Tansey KE, Theis JL, Tolfo CZ, Whitney M, Williams CD, Winter CM, Zanca JM. United States (US) multi-center study to assess the validity and reliability of the Spinal Cord Independence Measure (SCIM III). Spinal Cord. 2011 Aug;49(8):880-5. doi: 10.1038/sc.2011.20. Epub 2011 Mar 29. PMID 21445081